CLINICAL TRIAL: NCT00001295
Title: Continuing Treatment for Children and Adults in the Center for Cancer Research
Brief Title: Continuing Care and Treatment for Patients With Cancer/AIDS/Skin Disease
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920094; 92-C-0094
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-08-23

CONDITIONS: Cancer; HIV
Keywords: Follow-Up; Treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This protocol is to provide continuing medical/surgical/radio-therapeutic care, treatment and follow-up for NCI patients not currently entered on an active research protocol. No investigational treatments will be administered on this protocol.

DETAILED DESCRIPTION:
Background:

It may be in the interest of the CCR to continue to follow and treat certain subjects after they have completed their treatment and participation on a research protocol.

Objective:

To provide continuing treatment and medical follow-up for CCR subjects who have completed their treatment and participation on a research protocol and who are not currently entered on or eligible for another active research protocol.

Eligibility:

Subjects who have been previously enrolled on and received treatment according to an approved CCR research protocol. (clinical trial)

It is in the best interest of the subject and the CCR for the subject to continue to receive standard care and follow-up at the NIH.

Design:

Medical/surgical/radiotherapeutic care, treatment and follow-up is provided for CCR subjects who have completed their treatment and participation on a research protocol and who are not currently entered on an active research protocol.

No investigational treatments will be administered. This protocol is not be used as a platform to perform pilot studies of off-label uses for standard agents.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects of any age who have been previously enrolled and treated on an approved CCR research treatment protocol.

It is in the best interests of the subject and the CCR for the subject to continue to receive treatment and follow-up at the NIH.

The subject or guardian signs the informed consent and agrees to the proposed treatment regimen.

EXCLUSION CRITERIA:

Subjects who have not been previously treated on a CCR research treatment protocol.

Subjects who are receiving an investigational therapy.

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2145 (Actual)
Dates: Start 1992-01-29; Study Completion 2016-08-23

PRIMARY OUTCOMES:
To provide continuing treatment and medical follow-up for CCR subjects who have completed their treatment and participation on a research protocol and who are not currently entered on or eligible for an active research protocol. | Open-ended

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Steakley, R.N., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States